CLINICAL TRIAL: NCT04887038
Title: A Single and Multiple Dose-escalation First-in-human With Food-effect Study Evaluating the Safety, Tolerability and Pharmacokinetics of SRT-015 Administered Orally.
Brief Title: First-in-Human Study of SRT-015 in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SRT015-01
Record Dates: First submitted 2021-05-05; First posted 2021-05-14 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug :SRT-015 (Active Comparator): Experimental, Single and Multiple Oral escalating dose and Food Effect Cohort
  Interventions: Drug: SRT-015
- Matching Placebo for SRT-015 (Placebo Comparator)
  Interventions: Other: Matching Placebo for SRT-015

INTERVENTIONS:
Drug: SRT-015 — Each study part (A,B and C) will be completed sequentially, but with partial overlapping. The first cohort of Part B (Cohort B1) may be initiated after safety, tolerability and available PK data are assessed and deemed suitable to continue for a single dose on Part A that is equal to or greater than the total exposure of cohort B1. Part C (Cohort C1 & C2) may be initiated after safety, tolerability and PK data are assessed and deemed suitable to continue for a single dose in part A that is at least double the specified dose from part C.
  Arms: Drug :SRT-015
Other: Matching Placebo for SRT-015 — Matching Placebo
  Arms: Matching Placebo for SRT-015

SUMMARY:
This is phase 1 first-in-human trial evaluating SRT-015 to assess safety, tolerability and pharmacokinetics. This study will be conducted in 3 parts - SAD, MAD and Food Effect with target of 96 healthy volunteers.

This will be a single center, Phase 1, randomized, double-blind, placebo controlled, SAD and MAD study of dose escalation cohorts evaluating administration of SRT-015 or placebo. Additionally, PK will be assessed in fed and fasting states.

DETAILED DESCRIPTION:
The study will be divided into three parts:

Part A: SAD- Randomized, double-blind, placebo-controlled single oral escalating dose of SRT-015 or placebo in five cohorts (A1-A5). Each cohort will include 8 healthy subjects (6 randomized to receive SRT-015 and 2 to receive placebo). Two subjects from each cohort (1 to receive SRT-015 and 1 to receive placebo) will be dosed as sentinels, with the remainder of the subjects of each cohort (5 to receive SRT-015 and 1 to receive placebo) dosed at least the following day.

An extension cohort (Cohort A6) will allow investigation of a repeat or intermediate dose, at the discretion of the Sponsor or Safety Review Committee (SRC).

Part B: MAD- Randomized, double-blind, placebo-controlled multiple oral escalating dose of SRT-015 or placebo in four cohorts (B1-B4). Each cohort will include 8 healthy subjects (6 randomized to receive SRT-015 and 2 to receive placebo). Subjects will be treated with SRT-015 or placebo for 7 days.

An extension cohort (Cohort B5) will allow investigation of a repeat or intermediate dose at the discretion of Sponsor and SRC.

Part C: Food Effect (FE)- Randomized, crossover oral SRT-015 dose study of 8 healthy adults divided into two concurrent groups where half (n=4) of the subjects (Cohort C1) will receive the first dose as an oral suspension in fasting state on Day 1 of Period 1, the second dose as capsule formulation in fasting state on Day 1 of Period 2 and the third dose as a capsule formulation in a fed state on Day 1 of Period 3. The remainder (n=4) of the subjects (Cohort C2) will receive the first dose as an oral suspension in fasting state on Day 1 of Period 1, the second dose as a capsule formulation in a fed state on Day 1 of Period 2 and the third dose as a capsule formulation in a fasting state on Day 1 of Period 3.

ELIGIBILITY:
Key Inclusion Criteria:

1. Males or females aged 18 to 45 years of age with a BMI >18.0 and <32.0 kg/m2 and body weight greater than or equal to 50kg for males and greater than or equal to 45 kg for females.
2. Casual smoker (defined by the consumption of no more than 5 cigarettes per week, and willing to abstain from the consumption of cigarettes and related products for the study duration) or non smoker.
3. Agree to use appropriate contraception.

Key Exclusion Criteria:

1. Any clinically significant abnormality at physical examination, clinically significant abnormal laboratory test results (liver function tests must be strictly within normal ranges) or positive test for HIV, hepatitis B, or hepatitis C found during medical screening.
2. Positive urine drug screen or alcohol breath test at screening and check-in (Day -1).
3. Positive pregnancy test, or breast feeding.
4. Clinically significant 12-lead ECG abnormalities.
5. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability following of single and multiple oral doses of SRT-015 in healthy subjects | Up to two weeks
  Number of participants with serious and other non-serious adverse events
To evaluate the exposure to SRT-015 following single and multiple oral dose administration in healthy subjects (AUC last) | Up to two weeks
  Area under the serum concentration-time curve from time zero to last measurable concentration (mg*h/L)
3. To evaluate maximum serum concentration of SRT-015 following single and multiple oral dose administration in healthy subjects (Cmax) | Up to two weeks
  Maximum serum concentration (mg/L)

SECONDARY OUTCOMES:
To compare the exposure to SRT-015 (AUClast) in capsule formulation vs suspension formulation and fed vs fasted state | Up to two weeks
  Comparison of the area under the serum concentration-time curve from time zero to last measurable concentration after administration of SRT-015 after a meal v in a fasting state (mg*h/L)
To compare maximum serum concentration of SRT-015 (Cmax) in capsule formulation vs suspension formulation and fed v fasted state | Up to two weeks
  Maximum serum concentration (mg/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Pty Ltd, Victor Harbor, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No